CLINICAL TRIAL: NCT06279468
Title: Clinical Effectiveness of Intervertebral Disc Release in Treating Lenke 5 Adolescent Idiopathic Scoliosis (INDIRECT)
Brief Title: Clinical Effectiveness of Intervertebral Disc Release in Treating Lenke 5 Adolescent Idiopathic Scoliosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-23PJ2232
Record Dates: First submitted 2024-01-10; First posted 2024-02-28 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-02

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Intervertebral disc release; Adolescent idiopathic scoliosis; Derotation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IDR group (Experimental): A group designated as the IDR group will undergo subsequent intervertebral disc release following Ponte osteotomy on the predetermined vertebral levels.
  Interventions: Procedure: intervertebral disc release
- PO group (Active Comparator): The PO group will solely undergo Ponte osteotomy.
  Interventions: Procedure: Ponte osteotomy

INTERVENTIONS:
Procedure: intervertebral disc release — After standard posterior instrumentation and fusion in scoliosis cases, Ponte osteotomies are performed on vertebrae with a Nash-Moe classification of 1 degree or higher. The intervertebral discs on the convex side of the scoliosis, situated between the vertebrae that have undergone Ponte osteotomy, will be approached and incised parallel to the intervertebral space. The intervertebral disc and endplate cartilage were incised and separated using reamers. Subsequently, the intervertebral space was expanded and irrigated, and the fragments of the intervertebral disc were extracted using nucleus pulposus forceps. Impacting bone graft into the intervertebral space, thus sustaining the optimal height of intervertebral space.
  Other Names: IDR
  Arms: IDR group
Procedure: Ponte osteotomy — After standard posterior instrumentation and fusion in scoliosis cases, Ponte osteotomies are performed on vertebrae with a Nash-Moe classification of 1 degree or higher. Subsequent corrective procedures can be performed immediately following Ponte osteotomy completion. The deformity was corrected using the bilateral rod rotation and segmental derotation technique after inserting rods. Under fluoroscopic guidance, compression, distraction, and in situ bending maneuvers were implemented as needed. Allograft bone material was utilized for the purpose of bone fusion
  Other Names: PO
  Arms: PO group

SUMMARY:
Adolescent idiopathic scoliosis (AIS) poses challenges in achieving optimal three-dimensional correction. While posterior fusion with pedicle screws has shown success, osteotomy techniques, such as Ponte osteotomy, have further improved outcomes. However, residual vertebral rotation remains a concern, impacting long-term complications. Intervertebral disc release (IDR) presents a potential solution to enhance derotation and reduce fusion levels, particularly in Lenke Type 5 AIS. This prospective randomized controlled trial aims to evaluate the clinical effectiveness of IDR in treating Lenke 5 AIS, comparing it to Ponte osteotomy. The study focuses on axial vertebral rotation correction, coronal curve improvement, blood loss, hospital stay, and adverse events. Participants aged 10-18 with Lenke 5 AIS will undergo either IDR or Ponte osteotomy, randomly assigned. Outcome measures include axial rotation correction rate, radiographic parameters, and clinical assessments. A total of 132 participants will be recruited. The IDR technique, through posterior disc removal, presents a promising approach to optimize derotation in Lenke 5 AIS. While offering potential advantages, challenges like limited working space and bleeding risks require careful consideration. The study's findings aim to provide robust clinical evidence, enhancing treatment strategies for Lenke 5 AIS and offering innovative approaches for AIS as a whole.

DETAILED DESCRIPTION:
Hypotheses To examine the clinical effectiveness of intervertebral disc release in treating Lenke 5 adolescent idiopathic scoliosis, our working hypothesis posits that participants treated with intervertebral disc release achieve a higher rate of correction for axial vertebral rotation (especially the rotation of the apex vertebrae), demonstrate improved correction rate for coronal curve, experience no additional blood loss or allogeneic transfusions, and do not experience an increase in the length of hospital stay (LOH) or adverse event (AE) rate compared to individuals treated with Ponte osteotomy.

Objectives Based on the aforementioned hypothesis, this study aims to evaluate the clinical effectiveness of intervertebral disc release in treating Lenke 5 adolescent idiopathic scoliosis. The evaluation includes assessing the efficacy of vertebral derotation and the change in Cobb angle following the correction surgery, as well as perioperative blood loss, transfusion volume/rate, length of hospital stay, and the rate of adverse events (AEs).

Study setting and investigators The trial will take place at a tertiary care teaching hospital. The study will be conducted in the wards and operating rooms of the orthopedic department, which has 200 beds, at this comprehensive hospital with a total of 2500 beds. Participants will be recruited from the outpatient clinic by one investigator and will provide their consent to the investigators. All investigators have practical experience in clinical orthopedic research projects. A single team of surgeons, who have completed a clinical fellowship in spinal surgery, will perform the surgeries.

Participants The study will enroll patients between the ages of 10 and 18, with an American Society of Anesthesiologists (ASA) physical status classification of I-II. These patients will be diagnosed with Lenke 5 type adolescent idiopathic scoliosis and will require posterior correction, internal fixation, and bone graft fusion. Enrollment in the study will be contingent upon signing a written informed consent.

Patients with a history of previous corrective surgery, or with sharp, angulated short-segmental scoliosis, and those with congenital scoliosis requiring 3-column osteotomy will be excluded. Participants who experience dura mater laceration or unexpected massive bleeding during the operation will be excluded as well.

Randomization and concealment Before commencing the study, an independent researcher with no participant contact will utilize SAS 9.4 software (SPSS Inc., Chicago, IL, USA) to generate a blocked random number table (block size = 4). This table will be used to allocate eligible participants in a 1:1 ratio to 2 groups. A group designated as the IDR group will undergo subsequent intervertebral disc release following Ponte osteotomy on the predetermined vertebral levels, whereas the PO group will solely undergo Ponte osteotomy.

Data collection and monitoring The collected data will be entered into electronic case report forms (eCRFs) through a process of double data entry and logic validation. Subsequently, the eCRFs will be uploaded to a central server. To uphold the trial's quality standards, a proficient clinical trial expert will be invited to perform audits of both the trial implementation process and data entry on a bimonthly basis. The purpose of the regular audit is to ensure adherence to the protocol and Good Clinical Practices (GCPs). The expert may review source documents to verify the accuracy of the data recorded on CRFs. During each audit, all study records from the past 2 months will be thoroughly examined to ensure the quality of the trial conduct and the consistency between the source data and the data entered in the database. This study will not include any interim analysis.

Sample size and statistical analysis This trial will recruit 132 participants (66 participants per group) to confirm the primary outcome equivalence between IDR group and PO group. According to a prior study, the correction rate of axial rotation of the apex vertebrae is 0.60±0.23. Assuming that alpha = 0.05, power = 0.95, two-sided 95% CI, and the follow-up loss = 15%, 66 participants are needed for each group. G-power software version 3.1.9 was used for calculating the sample size. The primary outcome measures the correction rate of axial vertebral derotation. The mean values and standard deviations of these outcomes will be calculated for both the intervention and control groups. To assess the differences between the two groups, independent sample t-tests or Mann-Whitney U tests will be performed. Secondary outcomes measureå such as blood loss, allogeneic transfusions, length of hospital stay (LOH), and adverse events (AEs) will also be analyzed. Continuous variables (e.g., blood loss, LOH) will be analyzed using independent sample ttests or Mann-Whitney U tests, while categorical variables (e.g., allogeneic transfusions, AEs) will be analyzed using chi-square tests or Fisher's exact tests, as appropriate. The difference between the IDR group and PO group will be reported as mean difference and lower one-sided 95% confidence interval (CI), along with a one-sided p < 0.05. Statistical analyses will be conducted using SPSS.

Dissemination plan The trial results will be submitted to an international peer-reviewed journal. Additionally, the findings will be presented at relevant national and international conferences.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 10 and 18
* American Society of Anesthesiologists (ASA) physical statusclassification of I-II
* Lenke 5 type adolescent idiopathic scoliosis

Exclusion Criteria:

* A history of previous corrective surgery
* With sharp, angulated short-segmental scoliosis
* With congenital scoliosis requiring 3-column osteotomy

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
The correction rate of axial rotation of the apex vertebrae | immediately before surgery and one week after the surgery
  Axial rotation of apex vertebrae will be measured before and one week after the surgery using a novel computer-based automated measurement algorithm applied to computed tomography (CT) images. The algorithm used is a symmetry ratio algorithm that eliminates the need for manual landmark selection. It operates on the premise that the axis of maximum symmetry in a vertebral cross-section determines the angular orientation of the vertebra.

SECONDARY OUTCOMES:
Lumbar curve | immediately before surgery, 1-week post surgery, 3-month, 6-month, 1-year, 2-year, and 3-year follow-up
  the cobb angle of the lumbar curve
UIV tilt | immediately before surgery, 1-week post surgery, 3-month, 6-month, 1-year, 2-year, and 3-year follow-up
  the angle between the endplate of upper instrumented vertebra and the horizontal line
C7-CSVL | immediately before surgery, 1-week post surgery, 3-month, 6-month, 1-year, 2-year, and 3-year follow-up
  Radiographic parameters measured by CT scan: the distance between C7 vertebra and Central Sacral Vertical Line (CSVL)
Lumbar lordosis | immediately before surgery, 1-week post surgery, 3-month, 6-month, 1-year, 2-year, and 3-year follow-up
  the cobb angle of lumbar lordosis on sagittal plane
SVA | immediately before surgery, 1-week post surgery, 3-month, 6-month, 1-year, 2-year, and 3-year follow-up
  sagittal vertical axis, the distance between C7PL and CSVL
Radiographic parameters measured by CT scan: LIV and LIV+1 translation | immediately before surgery, 1-week post surgery, 3-month, 6-month, 1-year, 2-year, and 3-year follow-up
  the distance from the center of LIV or LIV+1 to CSVL
LIV tilt | immediately before surgery, 1-week post surgery, 3-month, 6-month, 1-year, 2-year, and 3-year follow-up
  the inclination in degrees of the inferior endplate relative to the horizontal
The lowest instrumented vertebra disc angle | immediately before surgery, 1-week post surgery, 3-month, 6-month, 1-year, 2-year, and 3-year follow-up
  the angulation in degrees between the inferior endplate of the LIV and the superior endplate of the next caudal vertebra
Age | immediately before surgery
  the age of patients
Gender | immediately before surgery
  the gender of patients
Risser grade of the patients at the time of surgery | immediately before surgery
  from 0 to 5, higher grades mean a worse outcome
number of fused spinal levels | immediately after surgery
  number of fused spinal levels in surgery
length of operation | immediately after surgery
  length of operation from incision to closure
Scoliosis Research Society-22,SRS-22 score | immediately before surgery, 1-week post surgery, 3-month, 6-month, 1-year, 2-year, and 3-year follow-up
  from 0 to 5, higher scores mean a better outcome
the MOS item short from health survey, SF-36 score | immediately before surgery, 1-week post surgery, 3-month, 6-month, 1-year, 2-year, and 3-year follow-up
  from 0 to 100, higher scores mean a better outcome
EuroQol Five Dimensions Questionnaire, EQ-5D score | immediately before surgery, 1-week post surgery, 3-month, 6-month, 1-year, 2-year, and 3-year follow-up
  from 0 to 5, higher scores mean a better outcome
Perioperative total blood loss | immediately after surgery
  Record perioperative total blood loss
Visible blood loss | immediately after surgery
  Record perioperative visible blood loss
Perioperative transfusion amounts | immediately after surgery
  Record perioperative transfusion amounts from treatment records
Perioperative transfusion rates | immediately after surgery
  Record perioperative transfusion rates from treatment records
Rate of postoperative infection | immediately after surgery
  Record the incidence rate of postoperative infection
The incidence of nerve damage | through study completion, an average of 3 years
  Record the incidence rate of nerve damage
The incidence of loss of correction | through study completion, an average of 3 years
  Record the incidence rate of loss of correction

CONTACTS AND LOCATIONS:
Overall Officials: Qianyu Zhuang, Professor, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No